CLINICAL TRIAL: NCT01759069
Title: The Effectiveness of a Microscope During Apical Surgery; a Prospective Randomized Controlled Clinical Trial.
Brief Title: RCT: Effectiveness of a Microscope During Dental Root Apical Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, M.H.T. de Ruiter, Resident/PhD student at dept. of Oral and Maxillofacial Surgery, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Microscope
Record Dates: First submitted 2012-12-24; First posted 2013-01-02 (Estimated); Last update posted 2014-01-20 (Estimated); Status verified 2014-01

CONDITIONS: Effectiveness of Microscope During Apical Surgery in Endodontic Treated Teeth.
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- treatment with microscope (Experimental): treatment with microscope
  Interventions: Procedure: Surgical treatment with microscope
- treatment without microscope (Experimental): treatment without microscope
  Interventions: Procedure: Surgical treatment with microscope

INTERVENTIONS:
Procedure: Surgical treatment with microscope

SUMMARY:
An endodontic treatment is the standard therapy for teeth with periapical periodontitis. The overall success rate for this treatment is high; 97% of the treated teeth are retained in the oral cavity after 8 years (Salehrabi & Rotstein, 2004). However, there are teeth that have a persistent granuloma because of various reasons and need endodontic retreatment or apical surgery. Overall results in literature for an endodontic retreatment show a success rate of 77%-89% (Ng, Mann, & Gulabivala, 2008; Salehrabi & Rotstein, 2010), the results of apical surgery are more or less similar (von Arx, 2005). Which of the two methods is preferred for failed root canal treatments is dependant on a variety of reasons. (For example an amount of gutta-percha outside the apex of the root is better corrected by apical surgery. Persistent infection as a result of insufficient gutta-percha amounts in a treated root is best treated with an endodontic retreatment.) The overall results in apical surgery have increased the past years due to better preparation of the apical end of the root by the use of an ultrasonic device (de Lange, Putters, Baas, & van Ingen, 2007) and new materials that are used for filling of the rootend e.g. MTA (von Arx, Hanni, & Jensen, 2010)

Objective of the study:

The objective of this study is to assess whether or not apical surgery that is carried out with the help of a microscope has a higher success rate than apical surgery without the use of a microscope. No RCT is found in present literature (Del Fabbro, Taschieri, Lodi, Banfi, & Weinstein, 2009).

ELIGIBILITY:
Inclusion Criteria:

* Peri-apical lesion on one of the teeth, confirmed on radiograph.
* Previous endodontic treatment was more than 6 months earlier.

Exclusion Criteria:

* Root fracture.
* Periodontal origin of apical infection or absence of marginal buccal bone after flap elevation.
* Root perforation.
* No previous endodontic treatment.
* Previous endodontic surgery.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2012-09; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Success is measured by Clinical outcome and radiographic assessment. | 6 months and 1 year
  A radiograph of the treated tooth is made directly post-operative, after 6 months and after 1 year post treatment. Clinical examination is performed at 6 months and 1 year after the operation.

CONTACTS AND LOCATIONS:
Locations (1):
- Academic Medical Center; Clinic of Oral and Maxillofacial Surgery, Amsterdam, Netherlands